CLINICAL TRIAL: NCT06207786
Title: Efficacy of Intranasal Povidone Iodine Swab Versus Oral Antibiotic Prophylaxis to Prevent Surgical Site Infections in Patients Undergoing Mohs Micrographic Surgery
Brief Title: Nasal Iodine Swab Versus Oral Antibiotic to Prevent Surgical Site Infection After Undergoing Mohs Micrographic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources to support the trial
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-009869
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Skin Cancer; Skin Cancer Face; Malignant Cutaneous Adnexal Neoplasm
MeSH Terms: conditions — Skin Neoplasms | interventions — Povidone-Iodine; Anti-Bacterial Agents; Amoxicillin; Azithromycin; Clarithromycin; Cephalexin; Clindamycin; Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: This randomized, open-label, single site clinical trial will be comprised of 2 comparison groups. Treatment arm 1 will be patients undergoing MMS for malignant cutaneous neoplasms receiving nasal povidone-iodine swabs prior to skin reconstruction. Treatment arm 2 will be patients undergoing MMS for malignant cutaneous neoplasms randomized to receive standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Povidone Iodine nasal swab (Experimental): Patients undergoing Mohs micrographic surgery (MMS) for malignant cutaneous neoplasms will receive nasal povidone-iodine swabs prior to skin reconstruction.
  Interventions: Other: Povidone-Iodine Swabs; Diagnostic Test: Staphylococcus nasal swab
- Oral antibiotic prophylaxis protocol (usual care) (Other): Patients undergoing Mohs micrographic surgery (MMS) for malignant cutaneous neoplasms will receive standard of care, including the provision of an oral anti-staphylococcal antibiotic per the standardized Antibiotic Prophylaxis protocol currently used for clinical decision making in Dermatologic Surgery at Mayo Clinic Rochester.
  Interventions: Diagnostic Test: Staphylococcus nasal swab; Drug: Antibiotic

INTERVENTIONS:
Other: Povidone-Iodine Swabs — Undergo nasal swab of both nostrils for 30 seconds into each nostril, allowing two minutes to dry, immediately (e.g. within 30 minutes) prior to performing skin reconstruction.
  Other Names: Betadine; Iodophore; Iodopovidone
  Arms: Povidone Iodine nasal swab
Diagnostic Test: Staphylococcus nasal swab — Undergo a nasal swab to identify patients with preoperative nasal Staphylococcus aureus colonization
Drug: Antibiotic — Receive an oral anti-staphylococcal antibiotic (e.g. oral cephalexin) with standard dosing only if indicated for antibiotic prophylaxis per the Mayo Clinic Dermatologic Surgery Antibiotic Prophylaxis protocol that is currently standard practice for patients undergoing Mohs micrographic surgery (MMS)
  Other Names: Amoxicillin; Azithromycin/clarithromycin; Cephalexin; Clindamycin; Trimethoprim-sulfamethoxazole
  Arms: Oral antibiotic prophylaxis protocol (usual care)

SUMMARY:
The purpose of this study is to compare surgical site infection rates for patients treated with Mohs micrographic surgery after bilateral nasal swab with povidone iodine versus standard treatment including the use of a standardized oral antibiotic prophylaxis protocol.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant, non-lactating/breastfeeding, non-incarcerated, English-speaking persons undergoing Mohs micrographic surgery (MMS) for malignant cutaneous neoplasms and receiving same-day defect repair by the MMS-performing surgeon
* Able to provide written informed consent prior to initiation of any study-specific procedures
* Able to swallow, retain, and absorb oral medications
* All malignant cutaneous neoplasms will be included

Exclusion Criteria:

* On antibiotic treatment or established intolerance or contraindication to povidone-iodine
* Allergy to specific oral antibiotics that are utilized as part of the Mayo Clinic Antibiotic Prophylaxis protocol (cefalexin, azithromycin, clindamycin)
* Requiring oral antibiotic therapy for prophylaxis postoperative infectious endocarditis or hematogenous total joint infection
* Cases where skin reconstruction is performed with non-sterile gloves
* Patients with lesions on the legs, as dilute vinegar soaks are standard practice and this would be a confounder for preventing surgical site infection
* Patients at increased risk for severe infections, including patients on immunosuppressive medications and biologics, patients with a history of HIV infection, chronic lymphocytic leukemia, immunodeficiency syndromes, as well as patients with insulin-dependent diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2029-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of nasal decolonization with povidone-iodine versus a standardized oral antibiotic prophylaxis protocol to prevent surgical site infection (SSI) | 30 days after MMS
  Effectiveness of nasal decolonization will be assessed based on the presence of SSI within 30 days after Mohs micrographic surgery (MMS). SSI is defined by the United States Centers for Disease Control and Prevention as infection of the cutaneous and subcutaneous tissue occurring within 30 days of surgery. Rates of SSI for both treatment arms will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Nahid Y. Vidal, M.D., Principal Investigator — Mayo Clinic in Rochester

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials